CLINICAL TRIAL: NCT04151173
Title: Assessment of Ovarian Reserve After Laparoscopic Cystectomy Versus Aspiration/Electrocoagulation in the Treatment of Ovarian Endometrioma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Collaborators: International Peace Maternity and Child Health Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiFMIH Jing Sun
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Ovarian Endometrioma; Ovarian Reserve
MeSH Terms: conditions — Endometriosis | interventions — Electrocoagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aspiration/electrocoagulation (Experimental)
  Interventions: Procedure: laparoscopic aspiration/electrocoagulation
- cystectomy (Active Comparator)
  Interventions: Procedure: laparoscopic cystectomy

INTERVENTIONS:
Procedure: laparoscopic aspiration/electrocoagulation — laparoscopic aspiration/electrocoagulation of ovarian endometrioma
  Arms: aspiration/electrocoagulation
Procedure: laparoscopic cystectomy — laparoscopic cystectomy of ovarian endometrioma
  Arms: cystectomy

SUMMARY:
This is a prospective, multicentric (three centers: 1: Shanghai First Maternity and Infant Hospital, Shanghai, China; 2: International Peace Maternity and Child Health Hospital, Shanghai, China, 3: Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai ,China), randomized clinical trial that includes patients undergoing laparoscopic surgery for primary unilateral ovarian endometriomas. Eligible patients will be subjected to transvaginal ultrasound before surgery to perform cyst classification (central type, marginal type and outcrop type). Patients are divided to two group: laparoscopic cystectomy group versus laparoscopic aspiration/electrocoagulation group. Biopsy samples in aspiration/electrocoagulation group and excision samples in cystectomy group are all subjected to histopathological examination. Follicular stimulating hormone (FSH), Anti mullerian hormone (AMH) and antral follicular count (AFC) will be measured pre-operative and post-operative.

The aim of the study is to determine whether and to what extent the two surgical procedures for ovarian endometrioma, cystectomy and aspiration/electrocoagulation, affect ovarian reserve. The investigators intend to confirm the clinical utility of ultrasonic classification of ovarian endometrioma, FSH, AMH and AFC in the assessment of ovarian reserve, and to promote their use in predicting decreased ovarian reserve.

The surgical excision of cystic wall, cystic fluid and peritoneal fluid will be subjected to transmission electron microscope, high resolution mass spectrometry and single-cell RNA sequencing to investigate their cellular and molecular features.

ELIGIBILITY:
Inclusion Criteria:

* Female with age between 18-40 years.
* Regular menstrual cycles
* Female diagnosed by ultrasound with unilateral ovarian endometrioma ≥4cm and ≤6cm.

Exclusion Criteria:

* Hormone, Gonadotropin-releasing hormone analogues or contraceptive therapy within 6 months before the current surgery and 6 months after surgery.
* Suspected or proven ovarian malignancy.
* Previous ovarian surgery.
* Evidence of polycystic ovary syndrome.
* Evidence of premature ovarian failure or premature menopause.
* Endocrinological diseases affecting ovarian reserve e.g. Diabetes mellitus, hypothyroidism.
* Pregnancy test is positive.
* Lactation.
* Unable or unwilling to give written consent.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
comparison between the impacts of laparoscopic cystectomy and laparoscopic aspiration /electrocoagulation on ovarian reserve as determined by alteration of AFC estimation in endometrioma patients. | 6 months
  AFC: number of follicles with average diameter of 2-10 mm in both ovaries assessed on day 2-5 of the menstrual cycle.

SECONDARY OUTCOMES:
comparison between the impacts of laparoscopic cystectomy and laparoscopic aspiration /electrocoagulation on ovarian reserve as determined by alteration of AMH level in endometrioma patients. | 6 months
  AMH is assessed on venous blood samples
comparison between the impacts of laparoscopic cystectomy and laparoscopic aspiration /electrocoagulation on ovarian reserve as determined by alteration of FSH level in endometrioma patients. | 6 months
  FSH is assessed on venous blood samples obtained on day 2-5 of the menstrual cycle

OTHER OUTCOMES:
Ultrasonic classification of ovarian endometrioma | Baseline (before laparoscopy)
  preoperative transvaginal ultrasonic classification of ovarian endometrioma (central type, marginal type and outcrop type)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality, China